CLINICAL TRIAL: NCT01048034
Title: Clinical and Biological Evaluation of Azacitidine in Transfusion-dependent Patients With Low and Intermediate-1 Risk MDS, and Low-risk CMML, Who Are Either Refractory to or Not Eligible for Treatment With Erythropoietin +/- G-CSF
Brief Title: Evaluation of Azacitidine in Transfusion Dependent Patients With Low-risk Myelodysplastic Syndrome (MDS) or Chronic Myelomonocytic Leukemia (CMML)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Nordic MDS Group (Network)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NMDSG08A; 2009-011483-11 (EudraCT Number)
Record Dates: First submitted 2010-01-12; First posted 2010-01-13 (Estimated); Last update posted 2013-10-29 (Estimated); Status verified 2013-10

CONDITIONS: Myelodysplastic Syndrome; Chronic Myelomonocytic Leukemia
Keywords: Myelodysplastic syndrome; Chronic myelomonocytic leukemia; Transfusion therapy; Transfusion dependency; Hypomethylating therapy; Azacitidine; DNA-methylation; Epigenetic modifications
MeSH Terms: conditions — Myelodysplastic Syndromes; Leukemia, Myelomonocytic, Chronic | interventions — Azacitidine; Erythropoietin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Azacitidine +/- erythropoetin (Experimental)
  Interventions: Drug: Azacitidine; Drug: Erythropoetin

INTERVENTIONS:
Drug: Azacitidine — 100 mg / m(2) subcutaneously day 1-5 every 4 weeks for 6 cycles. Another three cycles will be given together with epo for those not responding to the first 6 cycles of Azacitidine
Drug: Erythropoetin — For those patients not responding to Azacitidine alone, the combination of Azacitidine and erythropoetin 60 000 U / week for 16 weeks will be given.

SUMMARY:
Azacitidine has proved prolonged overall survival in patients with high-risk MDS. Minor pilot studies have shown that treatment with Azacitidine can induce transfusion independency in previous transfusion dependent patients with low-risk MDS. This study will evaluate the effect of Azacitidine in transfusion dependent patients with low-risk MDS (IPSS low or int-1) or low risk CMML. Included patients should first have failed, or considered not being eligible to, treatment with EPO +/- G-CSF. Our hypothesis is that Azacitidine can lead to transfusion independency in this group of patients. Those patients who do not respond to treatment with Azacitidine alone, will be given treatment with the combination of Azacitidine and EPO where our hypothesis is that Azacitidine can restore sensitivity to EPO.

ELIGIBILITY:
Inclusion Criteria:

* Must be 18 years of age at the time of signing the informed consent form
* MDS at IPSS Low or Int-1, or mixed MDS/MPD; either CMML with < 10% marrow blasts or RARS-T
* Patients with high or intermediate probability for response according to the predictive model (see Hellstrom-Lindberg et al, Br J Haematol 99:344-51 1997)should be refractory to EPO / darbepoetin (equivalent to > 60 000 U of EPO / week for > 8 weeks) followed by EPO + G-CSF for > 8 weeks, or biosimilar drugs in equipotent doses, or EPO + G-CSF upfront for 8 weeks. Patients with low probability for response according to the predictive model, could be included without prior EPO/G-CSF treatment
* Transfusion need >4 units over the last 8 weeks, or >8 units over the last 26 weeks.
* Subject has signed the informed consent document.
* Men and women of childbearing potential must use effective contraception during, and for up to 3 months after treatment.

Exclusion Criteria:

* Pregnant or lactating females.
* Patients who are eligible for curative treatment
* Expected survival less than 24 weeks.
* Symptomatic thrombocytopenia / active bleeding
* Patients with JAK-2 positive RARS-T if eligible for new investigational drugs
* Serum biochemical values as follows

  1. Serum creatinine >2.0 mg/dL (177 micromol/L)
  2. Serum aminotransferase (AST)/serum glutamic-oxaloacetic transaminase (SGOT) or alanine transaminase (ALT)/serum glutamate pyruvate transaminase (SGPT) >3.0 x upper limit of normal (ULN)
  3. Serum total bilirubin >1.5 mg/dL (26 micromol/L)
* Uncontrolled systemic infection
* Considered not capable of following the study protocol

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2010-01; Primary Completion 2012-08 (Actual); Study Completion 2012-08 (Actual)

PRIMARY OUTCOMES:
Hemoglobin level | Week 28
Number of patients reaching transfusion independency after treatment with Azacitidine | Week 28

SECONDARY OUTCOMES:
Effect on leucocyte, platelet count | Week 28 and End of Trial
Effect on bone marrow morphology and cytogenetics | Week 28 and End of Trial
Number of patients reaching transfusion independency after treatment with Azacitidine and Epo | End of Trial
Effect on genetic and epigenetic profile | Week 28
Hemoglobin level | End of Trial

CONTACTS AND LOCATIONS:
Overall Officials: Magnus Tobiasson, M.D., Study Director — Nordic MDS Group
Locations (17):
- Denmark (5):
  - Department of Hematology, Aalborg University Hospital, Aalborg
  - Department of Hematology, Aarhus Univsersity Hospital, Aarhus
  - Department of Hematology, Rigshospitalet Univsersity Hospital, Copenhagen
  - Department of Hematology, Herlev Hospital, Herlev
  - Department of Hematology, Odense University Hospital, Odense
- Norway (2):
  - Department of Medcine, Haukeland University Hospital, Bergen
  - Department of Hematology, Rikshospitalet University Hospital, Oslo
- Sweden (10):
  - Department of Medicine, Mälarsjukhuset Hospital, Eskilstuna
  - Department of medicine, Falun Hospital, Falun
  - Department of Medicine, Sahlgrenska University Hospital / Östra, Gothenburg
  - Department of Hematology, Linköping University Hospital, Linköping
  - Department of Medicine, Sunderbyn Hospital, Luleå
  - Department of Hematology, Lund University Hospital, Lund
  - Department of Hematology, Karolinska University Hospital, Stockholm
  - Department of Medicine, Södersjukhuset Hospital, Stockholm
  - Department of Medicine, Umeå University Hospital, Umeå
  - Department of Medicine, Uppsala University Hospital, Uppsala